CLINICAL TRIAL: NCT06944639
Title: Comparative Analysis of Three Types of Collagen Membranes Exposed to the Oral Environment: a Randomized Clinical Trial
Brief Title: Comparative Study of Three Collagen Membranes: 1 Non-cross-linked and 2 Cross-linked
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Ravida (Other)
Collaborators: Dentsply Sirona Inc. (Industry)
Responsible Party: Sponsor-Investigator, Andrea Ravida, Assistant Professor and Program director, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY24100119
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Bone Regeneration
Keywords: cross linked membrane; non cross linked membrane; degradation rate

STUDY DESIGN:
Intervention Model Description: All patients will receive the three membranes, placed randomly in different positions
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- OSSIX - BioMend - Jason (Active Comparator): Possible unique ordering of the 3 different membranes to which participants may be randomized
  Interventions: Device: Membrane Jason MB GmbH Non-cross-linked (NCL); Device: Membrane BioMend Extend Glutaraldehyde cross-linked; Device: Membrane OSSIX Agile Ribose cross-linked (RCL)
- BioMend - OSSIX - Jason (Active Comparator): Possible unique ordering of the 3 different membranes to which participants may be randomized
  Interventions: Device: Membrane Jason MB GmbH Non-cross-linked (NCL); Device: Membrane BioMend Extend Glutaraldehyde cross-linked; Device: Membrane OSSIX Agile Ribose cross-linked (RCL)
- BioMend - Jason - OSSIX (Active Comparator): Possible unique ordering of the 3 different membranes to which participants may be randomized
  Interventions: Device: Membrane Jason MB GmbH Non-cross-linked (NCL); Device: Membrane BioMend Extend Glutaraldehyde cross-linked; Device: Membrane OSSIX Agile Ribose cross-linked (RCL)
- Jason - OSSIX - BioMend (Active Comparator): Possible unique ordering of the 3 different membranes to which participants may be randomized
  Interventions: Device: Membrane Jason MB GmbH Non-cross-linked (NCL); Device: Membrane BioMend Extend Glutaraldehyde cross-linked; Device: Membrane OSSIX Agile Ribose cross-linked (RCL)
- Jason - BioMend - OSSIX (Active Comparator): Possible unique ordering of the 3 different membranes to which participants may be randomized
  Interventions: Device: Membrane Jason MB GmbH Non-cross-linked (NCL); Device: Membrane BioMend Extend Glutaraldehyde cross-linked; Device: Membrane OSSIX Agile Ribose cross-linked (RCL)
- OSSIX - Jason - BioMend (Active Comparator): Possible unique ordering of the 3 different membranes to which participants may be randomized
  Interventions: Device: Membrane Jason MB GmbH Non-cross-linked (NCL); Device: Membrane BioMend Extend Glutaraldehyde cross-linked; Device: Membrane OSSIX Agile Ribose cross-linked (RCL)

INTERVENTIONS:
Device: Membrane Jason MB GmbH Non-cross-linked (NCL) — The membrane will be stabilized in the oral mucosa using sutures and flowable composite.
Device: Membrane BioMend Extend Glutaraldehyde cross-linked — The membrane will be stabilized in the oral mucosa using sutures and flowable composite.
Device: Membrane OSSIX Agile Ribose cross-linked (RCL) — The membrane will be stabilized in the oral mucosa using sutures and flowable composite.

SUMMARY:
This study is being done to compare how quickly three different types of collagen membranes break down when they are exposed to the mouth. These membranes are often used in dental and oral surgery to help with healing and tissue growth. The goal is to find out if one membrane lasts longer than the others, which may help doctors choose the best option for different procedures.

In this study, the membranes will be placed in the mouth in a specific area near the gums of the upper back teeth. The study is designed so that neither the patients nor the researchers evaluating the results will know which membrane is which (this is called a double-blind study). Over time, researchers will measure how much each membrane has broken down. This information may help improve treatment planning and patient outcomes in dental care.

DETAILED DESCRIPTION:
The study was designed as a double-blinded, single-center, randomized clinical trial. Three different types of collagen membranes, ribose cross-linked (RCL) OSSIX Agile, glutaraldehyde cross-linked (GCL) - BioMend Extend, and non-cross-linked (NCL) Jason MB GmbH, were selected for the study.

During the first visit, digital intraoral impressions and clinical pictures will be taken, periodontal charts filled, and oral hygiene sessions conducted by trained hygienists. Two weeks later, during the second visit, patients will be reexamined to exclude any signs of inflammation. Membranes will be cut to a uniform size of 8*10 mm by an assistant prior to placement. They will be placed in a randomized mesiodistal order on the buccal mucosa, apical to the gingival margins of maxillary premolar and molar teeth (the future position will be evaluated on the intraoral scanned model). To fix the membranes, a vestibular sling suture without any perforation (PTFE 3/0) will be used. A light-cured periodontal dressing (Barricaid, Dentsply Caulk, Dentsply Int. Inc., York, PA, USA) will be placed on the buccal site to fix a knot and two other points on the membrane to fix it to the suture. Standard intraoral pictures will be taken. Patients will be instructed to avoid hard foods, brushing in the area of the membrane, and excessive movements to prevent dislocation of the structure. The same oral hygiene products will be provided to all patients.

Follow-up visits will be scheduled at 3, 7 and 10 days. At the 10-day follow-up clinical evaluation will be performed to assess any perforation. A set of pictures will be taken. Membranes integrity will be analyzed by two blinded examiners using a Scale.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Good overall health (ASA I or ASA II)
* Good oral health

Exclusion Criteria:

* Patients with gingival pathologies
* Individuals with uncontrolled chronic diseases or immunocompromised.
* Pregnant Patients
* Patients who are currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Degradation rates of three different collagen membranes simulating exposure to the oral environment. | 10 days
  Membrane integrity will be analyzed by two blinded examiners through photographs, using a scale from 0 to 5 where 0 means integrity and 5 represents complete resorption.

SECONDARY OUTCOMES:
Degradation rates of three different collagen membranes simulating exposure to the oral environment. | 3 and 7 days
  Membrane integrity will be analyzed by two blinded examiners through photographs, using a scale from 0 to 5 where 0 means integrity and 5 represents complete resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ravida, DDS, MS, PhD, Principal Investigator — Program Director of the Periodontics and Implant Dentistry Department
Locations (1):
- University of Pittsburgh, School of Dental Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klinger A, Asad R, Shapira L, Zubery Y. In vivo degradation of collagen barrier membranes exposed to the oral cavity. Clin Oral Implants Res. 2010 Aug;21(8):873-6. doi: 10.1111/j.1600-0501.2010.01921.x. PMID 20666799